CLINICAL TRIAL: NCT00785174
Title: Non-Invasive Ventilation Versus Continuous Positive Airway Pressure in Cardiogenic Pulmonary Edema: a Multicentre Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: President of Monastir University Tunisia, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIV-CPAP-CPE
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2008-11-05 (Estimated); Status verified 2008-11

CONDITIONS: Cardiogenic Pulmonary Edema
Keywords: noninvasive ventilation, continuous posi
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- continuous positive airway pressure (Active Comparator): respiratory assistance
  Interventions: Device: continuous positive airway pressure
- NIPSV (Active Comparator): respiratory assistance using face mak and ventilator to provide inspiratory pressure support and positive end expiratory pressure
  Interventions: Device: noninvasive pressure support ventilation

INTERVENTIONS:
Device: continuous positive airway pressure — respiratory assistance using face mask and positive expiratory pressure apllied by a Boussignac valve
  Other Names: Boussignac CPAP
  Arms: continuous positive airway pressure
Device: noninvasive pressure support ventilation — noninvasive pressure support ventilation can provide inspiratory pressure support and expiratory positive pressure
  Other Names: NIPSV
  Arms: NIPSV
Device: noninvasive pressure support ventilation — noninvasive pressure support ventilation provides an inspiratory aid and positive expiratory pressure using ventilator through face mask
  Other Names: NIPSV
  Arms: NIPSV

SUMMARY:
Non-invasive ventilation (NIV) has become now a widely used treatment modality in ICU and emergency services to deal with respiratory failure.1 NIV has the potential to improve ventilatory assistance while avoiding endotracheal intubation and its complications.

Since the first publications of Meduri2 and Brochard3 the number of studies on the NIV has been growing and developing and this technique becomes one of the major progress in the field of respiratory assistance. Decompensation of chronic obstructive pulmonary disease (COPD) is certainly the least questionable indication of the NIV. However, indication of the NIV is inexorably spreading to other types of acute respiratory insufficiency, including acute cardiogenic pulmonary edema (CPE).4 Continuous positive airway pressure (CPAP) is the most currently used non-invasive ventilation usually performed without the use of a ventilator. NIV using pressure support (NIPSV) combined pressure support (inspiratory aid) and positive expiratory pressure as in CPAP. Based on physiological ground, NIPSV would be more performant than CPAP to improve ventilatory parameters and reduce the work breathing in APE. However, this issue is not settled yet. Number of meta-analysis over the last 2 years were devoted to the comparison of CPAP and NISPV,5 so that the scientific evidence is still far from established. In addition, it is not sur that patients enrolled in these studies are representative of all patients with APE. The fact that they were included solely on the basis of clinical criteria, the risk of overlap with other diagnoses is not negligible. Thus the use of markers of heart failure as the BNP (brain natriuretic peptide) would be very useful. On the other hand, the possible deleterious effect of NIPSV on myocardial perfusion is a problem that has not been definitively resolved.

Objectives of the study:

1. Compare the efficacy and safety of the NIPSV with those of CPAP in patients presenting to the emergency department with CPE.
2. Compare the two procedures in subgroups of patients with hypercapnia and high BNP concentration.

DETAILED DESCRIPTION:
Cardiogenic pulmonary edema is defined as an increase of hydrostatic pressure in the pulmonary microcirculation resulting from postcapillaire hypertension.

The direct consequence is extravasation of fluid in the alveolar and interstitial tissue, leading to acute hypoxemia and a decrease in lung compliance. The decrease in lung compliance, increased airway resistance (interstitial and bronchial edema) and hypoxemia will cause an increase in work of breathing. The imbalance between the ability of respiratory muscles to generate effective gas exchange and exaggerated ventilatory load can lead to respiratory muscle fatigue requiring use of mechanical ventilation through endotracheal prosthesis. In addition, the increase in inspiratory muscles work during the CPE generates very important pleural depression, which increases transmural pressure and left ventricular afterload and thus increases pulmonary edema.

The CPAP is a non-invasive ventilation mode most currently used CPE. It is usually obtained via a mask and an expiratory valve to maintain constant pressure in the circuit. No inspiratory assistance is provided to the patient. The BOUSSIGNAC valve is currently used in clinical practice as an adjunct to the pharmacological treatment of CPE.The effect of CPAP is mainly linked to its ability to recruit zones that are collapsed during expiration. • NIPSV combines a positive expiratory pressure to ventilatory assistance pressure during inspiration delivered by a ventilator. It corresponds to a CPAP associated with inspiratory assistance, and thus, it is likely to improve the ventilation parameters, and in particular to reduce respiratory work more efficiently than CPAP alone.These beneficial physiological effects of NIPSV were well demonstrated during the decompensation of COPD ; they wait to be confirmed during CPE. Physiological studies have shown that the NIPSV is more effective in terms of reducing the work of breathing in CPE. However, none of the 7 published randomized studies has shown superiority of the NIPSV compared to CPAP in terms of reducing mortality and intubation requirement

ELIGIBILITY:
Inclusion Criteria:

* All patients aged >18 years and having acute respiratory failure caused by CPE.
* The origin of cardiogenic pulmonary edema is defined according to the history and clinical presentation, the chest X-ray and / or data of echocardiography when they are available with a serum BNP> 100pg/ml.

The acute respiratory failure is defined by the existence of clinical signs and / or arterial gas parameters:

* sweats and / or agitation and / or signs of struggle and /or drowsiness
* dyspnea with respiratory rate > 35/min,
* a blood oxygen saturation ≤ 90% by air.

Exclusion Criteria:

* Instability of the hemodynamic state (severe rhythm disturbances, hypotension with systolic arterial pressure <50 mmHg, need for inotropic drugs).
* The need for immediate endotracheal intubation.
* Contraindications to the use of a facial or nasal mask (or facial skin lesion).
* History of recent gastrointestinal surgery or pseudo obstruction.
* Refusal of participation or non-cooperation of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2005-01; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
It is the combination of 3 events: the need for endotracheal intubation, hospital death, and ICU hospitalisation. | 6 hours and 30 days after protocol start
Primary outcome It is the combination of 3 events: the need for endotracheal intubation, hospital death, and ICU hospitalisation. | 6 hours and 30 days after protocol start

SECONDARY OUTCOMES:
The change in the rate of troponin | 6 hours after protocol start
The length of hospital stay | 30 days after protocol start